CLINICAL TRIAL: NCT05418959
Title: Genetic Risk Stratification of Pediatric Skin Lesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elena Hawryluk, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022P001412
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Skin Lesion; Nevus
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Intervention Model Description: Non-invasive adhesive biopsies of suspicious skin lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DermTech PLA noninvasive adhesive biopsy (Experimental): Prior to surgical biopsy, a DermTech PLA noninvasive adhesive will be pressed over the lesion to collect superficial skin cells.
  Interventions: Diagnostic Test: DermTech PLA noninvasive adhesive biopsy

INTERVENTIONS:
Diagnostic Test: DermTech PLA noninvasive adhesive biopsy — The clinician will firmly press the DermTech noninvasive adhesive on the lesion and use their thumb to make five circular motions on the lesion. The adhesive patch will then be pulled off of the area. This will be repeated for an additional three patches.

SUMMARY:
A study to understand the clinical utility of noninvasive adhesive skin biopsies in pediatric patients by exploring whether DermTech Pigmented Lesion Assay (PLA) genetic risk analysis of suspicious lesions in children correlates with histopathological diagnosis.

DETAILED DESCRIPTION:
Patients (20 years of age or younger) with one or more atypical skin lesions requiring surgical biopsy within the next 6 months will be enrolled in the study. Prior to surgical biopsy, a DermTech PLA noninvasive adhesive will be performed on the lesion. The results of DermTech PLA genetic analysis will be compared to the results of histopathological diagnosis from surgical biopsy. Incidents of adverse events will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or younger.
* Subjects or parents willing and able to give informed consent, and assent as appropriate
* Patients will have one or more atypical skin lesions with management plan of monitoring, surgical biopsy, and/or excision of atypical nevi within the next 6 months

Exclusion Criteria:

* Lesions on palms, soles, mucosal membranes, or area where hair cannot be trimmed
* Bleeding or ulcerated lesions
* Previously biopsied, scarred, or known melanoma lesions
* Presence of active psoriasis/eczema/other skin condition in area to be biopsied

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of PRAME genetic marker. | 1 day
  Presence or absence of PRAME genetic marker from PLA test
Presence or absence of LINC genetic marker. | 1 da7
  Presence or absence of LINC genetic marker from PLA test

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 day
  No. of adverse events from adhesive skin biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Elena B Hawryluk, MD, PhD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jansen, B., Dobak, J. (2019) The Pigmented Lesion Assay Breakthrough: Enhanced Early Melanoma Detection with a Non-Invasive Gene Expression Test. DermTech, Inc. retrieved 4/11/20 from: https://dermtech.com/wp-content/uploads/PLA-TA.pdf
- [Background] Brouha B, Ferris LK, Skelsey MK, Peck G, Moy R, Yao Z, Jansen B. Real-World Utility of a Non-Invasive Gene Expression Test to Rule Out Primary Cutaneous Melanoma: A Large US Registry Study. J Drugs Dermatol. 2020 Mar 1;19(3):257-262. No abstract available. PMID 32550693